CLINICAL TRIAL: NCT06330961
Title: Effects of Different Kinds of Exercises in Pain, Lumbopelvic Biomechanics and Pain Pressure Thresholds in Patients With Non-specific Low Back Pain
Brief Title: Effects of Different Kinds of Exercise in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Daniel Sánchez-Zuriaga, Associate Professor, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023-MED-2756299
Record Dates: First submitted 2024-01-31; First posted 2024-03-26 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
Keywords: low back pain; isometric exercise; pain threshold; back muscles; surface electromyography
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain-free participants (Experimental): Aerobic exercise, Biering-Sorensen test and placebo interventions will be administered to a group of subjects with no past history of low back pain. They will serve as a control group.
  Interventions: Other: Isometric exercise; Other: Aerobic exercise; Other: Placebo intervention
- Low back pain patients (Experimental): Aerobic exercise, Biering-Sorensen test and placebo interventions will be administered to a group of non-specific low back pain patients. They will serve as the primary intervention group.
  Interventions: Other: Isometric exercise; Other: Aerobic exercise; Other: Placebo intervention

INTERVENTIONS:
Other: Isometric exercise — Biering-Sorensen maneuver.Participants will be in a prone position with the anterosuperior iliac spines on the edge of a stretcher. Their lower body will be strapped by the ankles and hips, with the upper body suspended. Participants will keep their trunk extended and parallel to the ground for 60 seconds.
Other: Aerobic exercise — After adjusting height, pedals and backrest in a cycloergometer, there will be 20 minutes of cycling, of which 5 minutes will be a warm-up at 50-60% of maximum heart rate and 15 minutes at 60-70% of maximum heart rate. There will be a constant monitoring of heart rate and oxygen saturation.
Other: Placebo intervention — A maneuver equivalent to Biering-Sorensen test, but with upper limb support on a level step and electromyographic monitoring to ensure minimal activation of the erector spinae. It will be explained to the participant that the aim of such an intervention is to cause electromyographic silence of the erector spinae and keep it for 1 minute.

SUMMARY:
Low back pain is considered one of the great global challenges in public health due to its high prevalence. Exercise have been shown to cause an increase in pain thresholds, through the effect known as exercise-induced hypoalgesia. Little is known about exercise-induced hypoalgesia induced by different modalities of exercise in low back pain, and its possible effects in lumbopelvic biomechanics.

The goal of this clinical trial is to compare the effect of exercise-induced hypoalgesia after an isometric, aerobic and a sham/ placebo exercise in non-specific low back pain. The main questions it aims to answer are:

* Does an isometric exercise intervention cause exercise-induced hypoalgesia in non-specific low back pain patients?
* Is the effect of an isometric exercise intervention comparable to that of aerobic exercise?
* Is a placebo/ sham intervention also effective to reduce pain thresholds in these patients?
* Do healthy subjects show the same effects in pain thresholds as low back pain patients ? Participants will perform an isometric, aerobic and placebo/ sham exercise intervention in three different recording sessions. Before and after the interventions, pain intensity, pain-pressure thresholds and lumbopelvic biomechanical parameters during trunk flexion-extension will be recorded.

Researchers will compare a group of low back pain patients to an age-, gender- and anthropometrics-matched control group of pain-free subjects to see if exercise-induced hypoalgesia is also observed when there is no low back pain diagnosis.

DETAILED DESCRIPTION:
Exercise causes an immediate reduction in pain sensitivity, known as exercise-induced hypoalgesia. This phenomenon is described as the immediate and lasting reduction of pain sensitivity after therapeutic exercise. This effect has been observed after isometric muscle contractions and aerobic exercises in healthy subjects.

The hypoalgesic response is often shown as an increase in pain-pressure thresholds in regions close to the most active muscle groups during exercise, and also in regions further away, which probably reflects the activation of systemic endogenous pain inhibitory systems. This effect has also been studied in patients with chronic pain.

Although there is previous work that has shown that aerobic exercise and isometric exercise can cause exercise-induced hypoalgesia, there is no evidence on exercise-induced hypoalgesia caused by isometric maneuvers in patients with low back pain. There is also a lack of placebo-controlled studies, or even studies comparing the analgesic effect of isometric and aerobic exercise in this population.

Therefore, the aim of this study will be to investigate, in a placebo-controlled intervention, whether various exercise modalities (isometric, aerobic) that involve activation of the lumbopelvic muscles result in local hypoalgesia in the area of the most active muscles, and/or hypoalgesia in more distant areas of the body, in subjects with low back pain and a group of healthy subjects which will serve as a control group.

ELIGIBILITY:
Inclusion Criteria:

Control group: no prior history of low back pain or any other kind of low back disorders.

Low back pain group:

* current symptoms of non-specific low back pain
* Symptoms must be severe enough to have caused recent loss of work days.

Exclusion Criteria:

* mental or cognitive impairment influencing the ability to understand and execute oral or written instructions
* any sign or symptom suggestive of potential underlying diseases
* presence of red flags or high-risk criteria for referral to emergency medical services
* severe functional limitation due to the intensity of the pain
* high irritability of symptoms at the time of the selection process
* inability to tolerate the prone position

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Day 1, before, after and 30 minutes past the first intervention. Day 8, before, after and 30 minutes past the second intervention. Day 15, before, after and 30 minutes past the third intervention.
  Pain intensity will be tested using a visual analogue scale, scored from 0 to 10.
Pain-pressure thresholds | Day 1, before, after and 30 minutes past the first intervention. Day 8, before, after and 30 minutes past the second intervention. Day 15, before, after and 30 minutes past the third intervention.
  Pain-pressure thresholds will be measured with an algometer on 3 points in a randomized order: 1) thenar eminence; 2) erector spinae (5 cm distal to L3); 3) the center of the long head of biceps femoris. Unit: kg/cm2
Trunk flexion-extension electromyography (EMG) | Day 1, before, after and 30 minutes past the first intervention. Day 8, before, after and 30 minutes past the second intervention. Day 15, before, after and 30 minutes past the third intervention.
  Average percentages of lumbopelvic muscles activation during flexion, extension, eccentric and concentric contractions and the myoelectrical silence, recorded by an EMG100C Biopac module (Biopac Systems, Inc., Goleta, CA). Unit: percentages of maximum muscle activation
Flexion-extension ratio (EMG) | Day 1, before, after and 30 minutes past the first intervention. Day 8, before, after and 30 minutes past the second intervention. Day 15, before, after and 30 minutes past the third intervention.
  A ratio between the average lumbopelvic muscles activity at trunk flexion and its average activity at extension, to quantify the relaxation level of the muscle. Unit: dimensionless
Maximum ranges of lumbar and pelvic flexion | Day 1, before, after and 30 minutes past the first intervention. Day 8, before, after and 30 minutes past the second intervention. Day 15, before, after and 30 minutes past the third intervention.
  Maximum ranges of lumbar and pelvic flexion, in degrees, measured with a Liberty 240/16 electrogoniometer (Polhemus Inc., Colchester, USA). Unit: degrees
Trunk flexion-extension percentages of motion | Day 1, before, after and 30 minutes past the first intervention. Day 8, before, after and 30 minutes past the second intervention. Day 15, before, after and 30 minutes past the third intervention.
  Average percentages of maximum lumbar and pelvic flexion during flexion and extension, and at the start and end of lumbopelvic muscles relaxation, measured with a Liberty 240/16 electrogoniometer (Polhemus Inc., Colchester, USA) and expressed as a percentage of the maximum range of flexion during each flexion-extension cycle. Unit: percentages of maximum flexion
Time of maximum flexion | Day 1, before, after and 30 minutes past the first intervention. Day 8, before, after and 30 minutes past the second intervention. Day 15, before, after and 30 minutes past the third intervention.
  Percentage of total flexion-extension time during which the lumbar spine and the pelvis are flexed over 90% of their maximum flexion, measured with a Liberty 240/16 electrogoniometer (Polhemus Inc., Colchester, USA). Unit: percentage of total flexion-extension time
Fear-avoidance beliefs | Day 1, before, after and 30 minutes past the first intervention. Day 8, before, after and 30 minutes past the second intervention. Day 15, before, after and 30 minutes past the third intervention.
  Fear-avoidance beliefs will be tested using a validated version of the Fear-Avoidance Beliefs Questionnaire (FABQ).
Pain distribution and supra-threshold stimulation | Day 1, before and after the first intervention. Day 8, before and after the second intervention. Day 15, before and after the third intervention.
  Area of pain irradiation, and area of distribution of pressure-induced referred pain after a supra-threshold stimulation over the infraspinatus muscle. Depicted by the participants on a body chart. Unit: cm2

SECONDARY OUTCOMES:
Anthropometric data: height | Day 1, before the first intervention. Day 8, before the second intervention. Day 15, before the third intervention.
  Measured with a stadiometer, barefoot. Unit: meters
Anthropometric data: weight | Day 1, before the first intervention. Day 8, before the second intervention. Day 15, before the third intervention.
  Measured with a calibrated scale with the participant barefoot and wearing light clothes. Unit: kilograms
Date of birth/ age | Day 1, before the first intervention.
  Self-reported. Unit: years
Sex/ gender | Day 1, before the first intervention.
  Self-reported
Basic clinical history and occupational data | Day 1, before the first intervention.
  Self-reported, in an interview. Antecedents of low back pain, occupation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sánchez-Zuriaga, PhD, MD, Principal Investigator — University of Valencia
Locations (1):
- Clinical Anatomy of the Musculoskeletal System Laboratory. Department of Anatomy and Human Embryology, School of Medicine, Universitat de València, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No